CLINICAL TRIAL: NCT04585646
Title: A Two-Week Crossover Dispensing Evaluation Of Orion Daily Wear Soft Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CV-20-18
Record Dates: First submitted 2020-10-05; First posted 2020-10-14 (Actual); Results first posted 2022-05-10 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-04

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Orion then Gemini (Experimental): Subjects will be randomized to wear Orion daily disposable contact lens then Gemini daily disposable contact lens for 2 weeks in this randomized, cross-over bilateral dispensing study.
  Interventions: Device: Orion daily disposable contact lens; Device: Gemini daily disposable contact lens
- Gemini then Orion (Experimental): Subjects will be randomized to wear Gemini daily disposable contact lens then Orion daily disposable contact lens for 2 weeks in this randomized, cross-over bilateral dispensing study.
  Interventions: Device: Orion daily disposable contact lens; Device: Gemini daily disposable contact lens

INTERVENTIONS:
Device: Orion daily disposable contact lens — Subjects will be randomized to wear Orion lens for 2 weeks.
Device: Gemini daily disposable contact lens — Subjects will be randomized to wear Gemini lens for 2 weeks.

SUMMARY:
The primary objective of the study is to evaluate the clinical performance of test lens (Orion) in comparison with control lens (Gemini) over a period of two weeks of wear.

DETAILED DESCRIPTION:
The primary objective of the study is to evaluate the clinical performance of test lens (Orion) in comparison with control lens (Gemini) over a period of two weeks of wear. This is a double-masked, randomized, bilateral, two-week crossover, dispensing study.

ELIGIBILITY:
Inclusion Criteria:

* Is at least 18 years of age and has full legal capacity to volunteer.
* Is no greater than 55 years of age.
* Has read and understood the information consent letter.
* Is willing and able to follow instructions and maintain the appointment schedule.
* Is an adapted soft contact lens wearer having worn lenses for a minimum of 4 weeks prior to the study.
* Has spectacle cylinder ≤1.00D in both eyes.
* Has spherical contact lens power requirement between -1.00D and -6.00D in both eyes.
* Has manifest refraction visual acuities (VA) equal to or better than logMAR equivalent of 20/20 in each eye.
* Wears CLs in both eyes (monovision acceptable, but not monofit)
* Has clear corneas and no active ocular disease.
* Has not worn lenses for at least 12 hours before the examination.
* Is willing to wear the study contact lenses for a minimum 8 hours per day/6 days per week

Exclusion Criteria:

* Has never worn contact lenses before.
* Has any systemic disease affecting ocular health.
* Is using any systemic or topical medications that will affect ocular health.
* Has any ocular pathology or severe insufficiency of lacrimal secretion (moderate to severe dry eyes) that would affect the wearing of contact lenses.
* Has persistent, clinically significant corneal or conjunctival staining using sodium fluorescein dye.
* Has any clinically significant lid or conjunctival abnormalities, active neovascularization or any central corneal scars.
* Is aphakic.
* Has strabismus/amblyopia.
* Has undergone corneal refractive surgery.
* Is pregnant, lactating or planning a pregnancy.
* Is participating in any concurrent clinical or research study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pete S Kollbaum, Principal Investigator — Indiana University
Locations (1):
- CORL, Indiana University, Bloomington, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Orion Then Gemini: Subjects were randomized to wear Orion daily disposable contact lens then Gemini daily disposable contact lens for 2 weeks in this randomized, cross-over bilateral dispensing study.
- Gemini Then Orion: Subjects were randomized to wear Gemini daily disposable contact lens then Orion daily disposable contact lens for 2 weeks in this randomized, cross-over bilateral dispensing study.
Period: First Intervention
Arm/Group | Orion Then Gemini | Gemini Then Orion
Started | 32 | 32
Completed | 31 | 28
Not Completed | 1 | 4
Not completed — Physician Decision | 1 | 0
Not completed — Lost to Follow-up | 0 | 3
Not completed — Withdrawal by Subject | 0 | 1
Period: Second Intervention
Arm/Group | Orion Then Gemini | Gemini Then Orion
Started | 31 | 28
Completed | 31 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Subjects were randomized to wear Orion daily disposable contact lenses for 2 weeks and then Gemini daily disposable contact lenses for 2 weeks in this randomized, cross-over bilateral dispensing study.
  Orion daily disposable contact lens Gemini daily disposable contact lens
Arm/Group | Overall Study
Number analyzed (Participants) | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 64
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 23 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 64

OUTCOME MEASURES:

1. Primary Outcome: Subjective Response for Vision Satisfaction
Description: Subjective Response for Vision Satisfaction assessed on 7-point Likert (Very satisfied, Satisfied, Somewhat satisfied, Neither Satisfied nor Dissatisfied, Somewhat Dissatisfied, Dissatisfied, Very Dissatisfied)
Time Frame: Baseline - After 10 minutes of lens dispense
Measure: Count of Participants; unit: Participants
Groups:
- Orion: Subjects were randomized to wear Orion daily disposable contact lenses for 2 weeks in this randomized, cross-over bilateral dispensing study.
  Orion daily disposable contact lens
- Gemini: Subjects were randomized to wear Gemini daily disposable contact lenses for 2 weeks in this randomized, cross-over bilateral dispensing study.
  Gemini daily disposable contact lens:
Arm/Group | Orion | Gemini
Number analyzed (Participants) | 59 | 59
Participants
  Very satisfied | 24 | 28
  Satisfied | 30 | 24
  Somewhat Satisfied | 4 | 7
  Neither | 1 | 0
  Somewhat Dissatisfied | 0 | 0
  Dissatisfied | 0 | 0
  Very Dissatisfied | 0 | 0

2. Primary Outcome: Subjective Response for Overall Vision Satisfaction
Description: as for outcome 1
Time Frame: 2 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Orion | Gemini
Number analyzed (Participants) | 59 | 59
Participants
  Very satisfied | 26 | 28
  Satisfied | 22 | 24
  Somewhat Satisfied | 7 | 5
  Neither | 0 | 1
  Somewhat Dissatisfied | 3 | 1
  Dissatisfied | 1 | 0
  Very Dissatisfied | 0 | 0

3. Primary Outcome: Subjective Response for Overall Vision Satisfaction
Description: as for outcome 1
Time Frame: 2 Weeks - at night
Measure: Number; unit: percentage of participants
Arm/Group | Orion | Gemini
Number analyzed (Participants) | 59 | 59
percentage of participants
  Very satisfied | 42 | 34
  Satisfied | 41 | 48
  Somewhat Satisfied | 8 | 10
  Neither | 7 | 3
  Somewhat Dissatisfied | 2 | 5
  Dissatisfied | 0 | 0
  Very Dissatisfied | 0 | 0

4. Primary Outcome: Subjective Response for Overall Vision Quality
Description: Subjective Response for Overall Vision quality assessed on a 0-100 scale (0- Unacceptable, 100- Excellent Vision)
Time Frame: Baseline - After 10 minutes of lens dispense
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Orion | Gemini
Number analyzed (Participants) | 59 | 59
units on a scale | 90 (8) | 91 (9)

5. Primary Outcome: Subjective Response for Overall Vision Quality
Description: Subjective Response for Overall Vision Quality assessed on a 0-100 scale (0- Unacceptable, 100- Excellent Vision)
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Orion | Gemini
Number analyzed (Participants) | 59 | 59
units on a scale | 86 (16) | 89 (10)

6. Primary Outcome: Subjective Response for Overall Vision Quality
Description: Subjective Response for Overall Vision Quality assessed on a 0-100 scale (0- Unacceptable, 100- Excellent Vision)
Time Frame: 2 weeks - Night Driving
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Orion | Gemini
Number analyzed (Participants) | 59 | 59
units on a scale | 87 (13) | 88 (10)

7. Secondary Outcome: Subjective Overall Comfort Satisfaction
Description: Overall comfort satisfaction analyzed on 7-point Likert (Very satisfied, Satisfied, Somewhat satisfied, Neither Satisfied nor Dissatisfied, Somewhat Dissatisfied, Dissatisfied, Very Dissatisfied)
Time Frame: Baseline - After 10 minutes of lens dispense
Measure: Count of Participants; unit: Participants
Arm/Group | Orion | Gemini
Number analyzed (Participants) | 59 | 59
Participants
  Very satisfied | 32 | 31
  Satisfied | 20 | 22
  Somewhat satisfied | 7 | 6
  Neither | 0 | 0
  Somewhat Dissatisfied | 0 | 0
  Dissatisfied | 0 | 0
  Very Dissatisfied | 0 | 0

8. Secondary Outcome: Subjective Overall Comfort Satisfaction
Description: as for outcome 7
Time Frame: 2 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Orion | Gemini
Number analyzed (Participants) | 59 | 59
Participants
  Very satisfied | 22 | 17
  Satisfied | 25 | 19
  Somewhat satisfied | 6 | 14
  Neither | 0 | 2
  Somewhat Dissatisfied | 4 | 4
  Dissatisfied | 2 | 3
  Very Dissatisfied | 0 | 0

9. Secondary Outcome: Subjective Preference for Comfort
Description: Subjective preference for comfort (Orion strongly, Orion slightly, No preference, Gemini slightly, Gemini strongly)
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 59
Participants
  Orion strongly | 13
  Orion slightly | 21
  No preference | 10
  Gemini slightly | 7
  Gemini strongly | 8

10. Secondary Outcome: Lens Surface Wettability Performance
Description: Lens Surface wettability performance was measured on a scale of 0-4, 0.25 steps (0-Very poor, 1 - Poor, 2- Acceptable, 3- Good, 4- Excellent)
Time Frame: Baseline - After 10 minutes of lens dispense
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Orion | Gemini
Number analyzed (Participants) | 59 | 59
units on a scale | 3.40 (0.36) | 3.32 (0.40)

11. Secondary Outcome: Lens Surface Wettability Performance
Description: as for outcome 10
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Orion | Gemini
Number analyzed (Participants) | 59 | 59
units on a scale | 3.31 (0.41) | 3.40 (0.38)

12. Secondary Outcome: Horizontal Lens Centration
Description: Horizontal Lens Centration assessed in primary gaze, white light, diffuse, low-medium magnification, with graticule on 0.1mm steps (Nasal decentration given +ve value. temporal decentration given -ve value)
Time Frame: Baseline - After 10 minutes of lens dispense
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Orion | Gemini
Number analyzed (Participants) | 59 | 59
mm | -0.12 (0.25) | -0.18 (0.26)

13. Secondary Outcome: Horizontal Lens Centration
Description: as for outcome 12
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Orion | Gemini
Number analyzed (Participants) | 59 | 59
mm | -0.13 (0.27) | -0.17 (0.27)

14. Secondary Outcome: Vertical Lens Centration
Description: Vertical Lens Centration assessed in primary gaze, white light, diffuse, low-medium magnification, with graticule on 0.1mm steps (Superior decentration given +ve value, inferior decentration given -ve value)
Time Frame: Baseline - After 10 minutes of lens dispense
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Orion | Gemini
Number analyzed (Participants) | 59 | 59
mm | 0.03 (27) | 0.06 (0.29)

15. Secondary Outcome: Vertical Lens Centration
Description: as for outcome 14
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Orion | Gemini
Number analyzed (Participants) | 59 | 59
mm | 0.09 (0.27) | 0.12 (0.32)

16. Secondary Outcome: Post-blink Movement
Description: Post-blink movement assessed on the amount of lens movement to the nearest 0.1mm immediately after the blink
Time Frame: Baseline - after 10 minutes of lens dispense
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Orion | Gemini
Number analyzed (Participants) | 59 | 59
mm | 0.28 (0.08) | 0.29 (0.09)

17. Secondary Outcome: Post-blink Movement
Description: Post-blink movement assessed on the amount of lens movement to the nearest 0.1mm immediately after the blink
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Orion | Gemini
Number analyzed (Participants) | 59 | 59
mm | 0.29 (0.08) | 0.32 (0.09)

18. Secondary Outcome: Lens Horizontal Mobility Rating
Description: Lens Horizontal Mobility Rating on a scale of 0-4 (0-immobile, 1- restricted, 2- secure, 3- unrestricted, 4- very mobile)
Time Frame: Baseline - after 10 minutes of lens dispense
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Orion | Gemini
Number analyzed (Participants) | 59 | 59
units on a scale | 2.36 (0.30) | 2.33 (0.29)

19. Secondary Outcome: Lens Horizontal Mobility Rating
Description: as for outcome 18
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Orion | Gemini
Number analyzed (Participants) | 59 | 59
units on a scale | 2.36 (0.28) | 2.41 (0.31)

20. Secondary Outcome: Corneal Staining Extent
Description: Corneal staining extent will be assessed on a scale of 0-4 (0- No Staining, 1- 1 to 15% of area, 2- 16 to 30% of area, 3- 31-45% of area, 4- >45% of area).
Time Frame: Baseline - after 10 minutes of lens dispense
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Orion | Gemini
Number analyzed (Participants) | 59 | 59
units on a scale
  Central | 0.00 (0.00) | 0.00 (0.00)
  Nasal | 0.01 (0.09) | 0.01 (0.09)
  Temporal | 000 (0.00) | 0.00 (0.00)
  Superior | 0.00 (0.00) | 0.00 (0.00)
  Inferior | 0.01 (0.09) | 0.01 (0.09)

21. Secondary Outcome: Corneal Staining Extent
Description: as for outcome 20
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Orion | Gemini
Number analyzed (Participants) | 59 | 59
units on a scale
  Central | 0.00 (0.00) | 0.00 (0.00)
  Nasal | 0.02 (0.13) | 0.01 (0.09)
  Temporal | 0.00 (0.00) | 0.00 (0.00)
  Superior | 0.00 (0.00) | 0.00 (0.00)
  Inferior | 0.01 (0.38) | 0.15 (0.39)

22. Secondary Outcome: Overall Lens Fit Acceptance
Description: Overall Lens Fit Acceptance assessed on a scale of 0-4 (0-Can't be worn, 1- Poor but acceptable, 2- Fair, 3- Good, 4- Optimum)
Time Frame: Baseline - after 10 minutes of lens dispense
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Orion | Gemini
Number analyzed (Participants) | 59 | 59
units on a scale | 3.20 (0.32) | 3.11 (0.32)

23. Secondary Outcome: Overall Lens Fit Acceptance
Description: as for outcome 22
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Orion | Gemini
Number analyzed (Participants) | 59 | 59
units on a scale | 3.22 (0.34) | 3.11 (0.39)

24. Secondary Outcome: Lens Handling Satisfaction
Description: Lens handling satisfaction assessed on a 7-point Likert Scales (Very satisfied, satisfied, Somewhat satisfied, Neither Satisfied nor Dissatisfied, Somewhat Dissatisfied, Dissatisfied, Very Dissatisfied)
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Orion | Gemini
Number analyzed (Participants) | 59 | 59
Participants
  Very satisfied | 27 | 14
  satisfied | 20 | 27
  Somewhat satisfied | 8 | 11
  Neither | 2 | 3
  Somewhat Dissatisfied | 1 | 3
  Dissatisfied | 1 | 1
  Very Dissatisfied | 0 | 0

25. Secondary Outcome: Subjective Overall Lens Handling
Description: SubjectiveOverall Lens handling assessed on a scale of 0-100 (0- cannot be managed, 100- Excellent handling)
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Orion | Gemini
Number analyzed (Participants) | 59 | 59
units on a scale | 87 (14) | 83 (16)

ADVERSE EVENTS:
Time Frame: From dispense up to 2 weeks on each study lens, a total of 4 weeks,
Arm/Group | Orion | Gemini
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/64
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/64
Other Adverse Events (participants affected / at risk) | 0/64 | 0/64

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-20): https://cdn.clinicaltrials.gov/large-docs/46/NCT04585646/Prot_SAP_000.pdf